CLINICAL TRIAL: NCT01886391
Title: Health Behavior-Related Outcomes With Diaphragmatic Breathing Retraining in Heart Failure Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Major changes in study required new IRB application and approval
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0179-09-FB; 5P20NR011404-03 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; Dyspnea; Diaphragmatic breathing retraining; Fatigue; Health-related Outcomes
MeSH Terms: conditions — Heart Failure; Dyspnea; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diaphragmatic Breathing Retraining (Experimental): Diaphragmatic breathing retraining (DBR) with a slow breathing pattern such that breathe in slowly through the nose for 4 seconds and breathe out slowly through the mouth for 6 seconds and mediated by Self-efficacy for DBR. Patients in this group will receive detailed instructions, in-person, as to how to carry out the DBR intervention at home. They will provide a return demonstration to the research staff about how to do the deep breathing. They will also receive a written script of the DBR intervention. In addition to the script, patients in this group will receive 3 audio CDs (1 for week 1 [5-min DBR], 1 for week 2 [10-min DBR], 1 for weeks 3-8 [15-min DBR]), developed by the PI, to use to practice their deep breathing.
  Interventions: Behavioral: Diaphragmatic Breathing Retraining

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing Retraining — Diaphragmatic breathing retraining (DBR) with a slow breathing pattern such that breathe in slowly through the nose for 4 seconds and breathe out slowly through the mouth for 6 seconds and mediated by Self-efficacy for DBR. Patients in this group will receive detailed instructions, in-person, as to how to carry out the DBR intervention at home. They will provide a return demonstration to the research staff about how to do the deep breathing. They will also receive a written script of the DBR intervention. In addition to the script, patients in this group will receive 3 audio CDs (1 for week 1 [5-min DBR], 1 for week 2 [10-min DBR], 1 for weeks 3-8 [15-min DBR]), developed by the PI, to use to practice their deep breathing.

SUMMARY:
The purpose of this study is to provide information on how the practicing of deep breathing ("DBR" - diaphragmatic breathing re-training) may improve the health outcomes and likelihood of heart failure patients to engage in health-promoting activities by successfully controlling their shortness of breath (dyspnea).

DETAILED DESCRIPTION:
In heart failure (HF) patients, dyspnea (shortness of breath), a key contributor to and the strongest predictor of a chief reason for hospital readmission with fatigue, are the primary reasons for modification in function leading to decreased physical activity (PA). Dyspnea and fatigue lead to activity avoidance, subsequent muscle de-conditioning, and further increases of dyspnea at even lower levels of activity. Depression, because of its moderate relationship both with perceived functional status and dyspnea, can further diminish PA and increase disability in activities of daily living (ADLs). Strategies to minimize or mitigate dyspnea and to boost motivation are imperative for improving adherence to PA, and, in turn, improving fatigue, muscle weakness, PA itself, functional status, disability, and depression in HF patients. Thus, diaphragmatic breathing retraining (DBR) or deep breathing with a slow breathing pattern, a focus on decreasing dyspnea, and mediated by Self-efficacy for DBR and informal caregiver support during the DBR provide an innovative approach to positively impact the spiraling effects of HF. The purpose of this pilot/feasibility study is to evaluate a diaphragmatic breathing retraining (DBR) intervention that incorporates informal caregiver coaching to improve the primary outcomes of dyspnea, fatigue, and muscle weakness, and the secondary outcomes of PA, functional status, depression, disability, and depression.

ELIGIBILITY:
Inclusion Criteria:

* adults age 19 or older who have Class III through IV heart failure as classified by the New York Heart Association (NYHA)
* cognitively intact indicated by being able to describe what participation in the study will involve
* have a consistent informal caregiver, who is willing to provide support to the participants, and a telephone
* residing in a rural area (population less than 2,500) (U.S. Census, 1995).

Exclusion Criteria:

* myocardial infarction or coronary bypass surgery within the last three months
* active chest pain
* uncontrolled arrhythmia (atrial fibrillation or ventricular tachycardia)
* on transplant list or has ventricular assist device
* skeletal or neurological conditions that would impact muscle strength or interfere with 6 minute walk test (6MWT) (amputation, severe arthritis, Parkinson's, stroke, or severe neuropathy)
* history of severe COPD.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-05-15 (Actual); Study Completion 2012-05-15 (Actual)

PRIMARY OUTCOMES:
Effect of deep breathing to control shortness of breath and fatigue by slowing breathing to 6 breaths per minute. | baseline, after 8 week intervention and 3 months after 8 week intervention
  Dyspnea is measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) and by 18 items of dyspnea from activities composed of basic activities of daily living (ADLs), instrumental activities of daily living (IADLs), and other activities related to physical functioning using a 10-point Liker scale. Fatigue will be measured by 8-items from the PROMIS-57 Profile v.10.

SECONDARY OUTCOMES:
Effect of deep breathing on the secondary outcomes of muscle strength, physical activity, functional status, disability in activities of daily living, and instrumental activities daily living, depression, and quality of life. | baseline, after 8 week intervention and 3 months after 8 week intervention
  Muscle strength is measured by Nicholas dynamometer (Model 01160, Lafayette Instrument Co., Lafayette, IN). Physical activity is measured by 7-items from Behavioral Risk Factor Surveillance System (BRFSS) (BRFSS, 2009; Kohl & Kimsey, 2009), ActiHeart (Respironics, Inc.), and ActiGraph (Model GT3X, Pensacola, FL). Functional status is measured by 6-MWT and Timed Get Up & Go. Disability in ADLs & IADLs is measured by restriction & modification in performance of 13 activities composed of basic ADLs (bathing, dressing, feeding, transfer, continence, & toilet) & IADLs (shopping, transportation, telephone, preparing meals, housework, taking medication, and handling money) taken from the Older American Resource Services (OARS) tool. Depression is assessed by 21-item Beck Depression Inventory II (Beck et al., 1996) using a 4-point Likert scale. Quality of life is measured by the EuroQol 5-D (EQ-5D; The EuroQol Group, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Yaewon Seo, PhD, RN, Principal Investigator — University of Nebraska; Bernice Yates, PhD, RN, Study Director — University of Nebraska